CLINICAL TRIAL: NCT06939959
Title: Evaluating the Efficacy of Topical Insulin for the Restoration of Ocular Surface Interface in Dry Eye Disease.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Shafiq Tanveer, Resident Ophthalmologist, Khyber Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 579/DME/KMC
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Dry Eye; Insulin Sensitivity
Keywords: DRY EYE DISEASE; Topical Insulin; Ocular Surface Interface restoration
MeSH Terms: conditions — Dry Eye Syndromes; Insulin Resistance | interventions — Lubricant Eye Drops; Insulin

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial for the treatment of dry eye disease with two arms: topical artificial tears and topical insulin.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients will be masked for the treatment, but not the principle investigator. Another investigator will prepare the topical insulin according to a written protocol. Participants will be given a white, unlabeled eye dropper containing the same volume of artificial tears or topical insulin for groups I and II respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participant Group/Arm (Placebo Comparator): Artificial tears Artificial tears 4 times a day
  Interventions: Drug: Artificial tear
- Intervention Group/Arm (Experimental): Experimental: Insulin Topical insulin 1UI/ml 4 times a day
  Interventions: Drug: insulin human

INTERVENTIONS:
Drug: Artificial tear — commercially available artificial tears will be used consisting of same ingredients.
  Other Names: ARTIFICIAL TEARS
  Arms: Participant Group/Arm
Drug: insulin human — injection humulin will be used to make topical insulin drops
  Other Names: HUMULIN INSULIN
  Arms: Intervention Group/Arm

SUMMARY:
This is a parallel randomized controlled trial for the treatment of dry eye disease. The main objective is to investigate the efficacy and safety of the use of insulin eye drops in the control of moderate-severe dry eye disease. Topical insulin drops will be compared to artificial tears in improving the ocular surface interface in patients with dry eye disease over 1 year period.

DETAILED DESCRIPTION:
Patients fulfilling the selection criteria will be enrolled from eye OPD of KTH. A written informed consent will be taken after explaining the purpose of study. Data will be collected on a pre-designed structured proforma. Demographic data including age, gender, educational status, socioeconomic status will be noted. Each participant will undergo a complete history assessment and the OSDI score will be calculated after taking extensive history. Ophthalmologic examination, including visual acuity, refraction, slit-lamp examination, corneal staining, schirmer test and TBUT will be performed in each patient. Both eyes will be selected for each secondary outcome measure (TBUT & SCHIRMER TEST). However, only one OSDI score could only be obtained per patient for assessing primary outcome. All the previous medications used for dry eye will be stopped Participants' eyes will be randomized by blocked randomization in a 1:1 ratio to be treated with topical artificial tears (group I) and topical insulin 1U/ml (group II). The patients will be masked for the treatment, but not the principle investigator. Another investigator will prepare the topical insulin according to a written protocol. Participants will be given a white, unlabeled eye dropper containing the same volume of artificial tears or topical insulin for groups I and II respectively. Group I will receive artificial tears (control group) four times daily. Group II will receive topical insulin of 1u/ml four times daily. Follow-up assessments will be conducted at 4, 8 and 12 weeks for each participant to measure changes in TBUT, schirmer test, and OSDI score.

ELIGIBILITY:
Inclusion Criteria:

* Patients having Schirmer's test values of less than 10mm after 5 minutes of the procedure recording plus a non-invasive tear breakup time (TBUT) of less than 10 seconds and the Ocular Surface Disease Index (OSDI) of more than 32 (diagnosed as dry eye disease as per the operational definition of this study).
* any gender.
* aged 18 years and above.

Exclusion Criteria:

* Patients with active ocular infection, severe ocular surface disease other than Dry eye disease, and those who have undergone ocular surgery within the past 6 months.
* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
OSDI Score | 12 weeks or 3 months
  The treatment will be deemed effective if OSDI score of less than 20 is achieved at 12 weeks of the initiation of treatment

SECONDARY OUTCOMES:
TBUT & SCHIRMER TEST | 12 weeks or 3 months
  The treatment will be deemed effective if Schirmer's test values are above 10mm after 5 minutes, TBUT of more than 10 seconds s achieved at 12 weeks of the initiation of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shafiq Tanvee, MBBS, FCPS, Principal Investigator — KHYBER TEACHING HOSPITAL PESHAWAR KPK PAKISTAN
Locations (1):
- Khyber Teaching Hospital, Peshawar, Khyber Pukhtunkhwa, Pakistan

REFERENCES:
- [Background] Kawahara A. Treatment of Dry Eye Disease (DED) in Asia: Strategies for Short Tear Film Breakup Time-Type DED. Pharmaceutics. 2023 Nov 5;15(11):2591. doi: 10.3390/pharmaceutics15112591. PMID 38004570
- [Background] Zhang X, Zhao L, Deng S, Sun X, Wang N. Dry Eye Syndrome in Patients with Diabetes Mellitus: Prevalence, Etiology, and Clinical Characteristics. J Ophthalmol. 2016;2016:8201053. doi: 10.1155/2016/8201053. Epub 2016 Apr 26. PMID 27213053
- [Background] Aniah Azmi N, Bastion MC. Short-Term Results of Trial of Topical Insulin for Treatment of Dry Eyes in Diabetics. Eye Contact Lens. 2020 Jan;46 Suppl 1:S25-S32. doi: 10.1097/ICL.0000000000000623. PMID 31145207
- [Background] Tahmaz V, Menghesha L, Stern ME, Holtick U, Scheid C, Steven P. Insulin eye drops for severe refractory chronic ocular graft-versus-host disease. Bone Marrow Transplant. 2024 Jul;59(7):1031-1033. doi: 10.1038/s41409-024-02272-9. Epub 2024 Apr 10. No abstract available. PMID 38600163
- [Result] Markoulli M, Hui A. Emerging targets of inflammation and tear secretion in dry eye disease. Drug Discov Today. 2019 Aug;24(8):1427-1432. doi: 10.1016/j.drudis.2019.02.006. Epub 2019 Feb 22. PMID 30802601